CLINICAL TRIAL: NCT06222047
Title: The Effect of Breast Milk and Dextrose on the Orogastric Tube Insertion-related Pain and Comfort Levels of Preterm Babies
Brief Title: Pain and Comfort Level During Orogastric Catheter Insertion in Preterms
Acronym: OGpreterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., RN, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: buchOG
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Prematurity; Pain Acute; Comfort; Orogastric Tube Insertion
MeSH Terms: conditions — Premature Birth; Acute Pain | interventions — Milk, Human; Glucose

STUDY DESIGN:
Intervention Model Description: Breast Milk Dextrose Control
Who Masked: Outcomes Assessor
Masking Description: Breast milk and dextrose video recording It was applied just before starting. It is not clear which intervention was made before the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast milk (Experimental): Breast Milk Intervention: Wrapping was applied to the baby as a standard approach. 2 minutes before the insertion of the oragastric catheter, 2 ml of breast milk was given to the babys mouth with a syringe. After the baby was given breast milk, video recording started. The steps for inserting an orogastric catheter were followed, and the baby was monitored in an incubator during the application, with pulse and saturation monitored.
  Interventions: Other: breast milk
- Dextrose (Experimental): Dextrose Intervention: The baby will receive wrapping as standard treatment. The orogastric catheter is visible to the brim with 2 ml of 20% dextrose syringe 2 minutes before the insertion chamber (Bueno et al., 2013). After the baby is given dextrose, the video recording will start. The steps of the orogastric tube insertion procedure will be followed. The baby will be in an incubator during the application, with pulse and saturation monitored.
  Interventions: Other: dextrose
- Control group (No Intervention): The control group: Baby will be wrapped as standard treatment. Video recording will start 2 minutes before the baby is inserted into the orogastric catheter. The steps of the orogastric tube insertion procedure will be followed. The baby will be in an incubator during the application, with pulse and saturation monitored. No additional intervention will be applied to the baby.

INTERVENTIONS:
Other: breast milk — give breast milk before the OG catheter insertion
  Arms: Breast milk
Other: dextrose — give %20 dextrose before the OG catheter insertion
  Arms: Dextrose

SUMMARY:
Purpose of the research:

This research was planned to evaluate the effect of breast milk and dextrose application, which are pain relief methods, on the pain and comfort levels of preterm babies who will have an orogastric tube inserted in the 3rd and 4th levels of the Neonatal Intensive Care Unit.

Hypotheses:

H0: The methods used during orogastric tube insertion do not affect the pain and comfort levels of preterm babies.

H1: Preterm babies who are breastfed feel less pain during orogastric tube insertion.

H2: Preterm babies given dextrose during orogastric tube insertion feel less pain.

H3: The comfort level of preterm babies who are breastfed during orogastric tube insertion is higher.

H4: The comfort level of preterm babies given dextrose during orogastric tube insertion is higher.

H5: There is a difference between the pain and comfort levels of preterm patients in terms of group, time, and group-time, depending on the intervention applied.

DETAILED DESCRIPTION:
The orogastric will then be informed about the investigations of the premature babies to be removed. It will be held in a place where video recordings will be taken from the parent during the orogastric catheter insertion process. After informed consent is obtained, the group to be included will be determined by predetermined stratified randomization.

Standard treatment will be applied to all preterms. Standard approach; Wrapping data during painful and stressful interventions is an effective method to calm the data and shorten the spread (Gardner and Goldson, 2011). As shown by Erkut and Yıldız with 74 newborns, births wrapped during heel bleeding had lower pain scores and higher oxygen saturation temperatures than the control groups (Erkut and Yıldız, 2017). The wrapping application will be wrapped in the flexion and abduction positions of the pre-terms, as a subscription for all members, in a way that does not cause movement restriction.

Babies are cared for every morning between 08.00 and 08.30. During care, orogastric catheters, tubes, and probes are renewed. Hand, face, and body care and oral care are provided and diapers are changed. Orgastric catheters of the babies included in the study will be removed during care hours. Maintenance takes approximately 15 minutes. Wrapping will be applied as standard treatment to all babies included in the study. After the care was done, it was wrapped early and allowed to rest. They are fed at 09.00. Preterms to be included in the study in each group; 30-45 without insertion of orogastric tube. They will be wrapped up in their beds and will be in a rest period where they will not be disturbed until minutes before. Oragastric catheters will be removed before feeding at 9:00. Video recording will be made starting before the procedure of connecting to the oragastric catheter (2 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Birth week 32-34,

  * Postnatal week has reached 32-34 weeks,
  * Birth weight over 1500 grams,
  * whose general condition is stable,
  * Planned to insert an orogastric tube,
  * Developed sucking and swallowing reflexes, being able to hold a pacifier,
  * Having breast milk,
  * Preterms whose parents agreed to participate in the study were included in the study.

Exclusion Criteria:

* In need of oxygen support,

  * Receiving analgesic and/or sedation treatment,
  * In the preoperative and/or postoperative period,
  * Those with congenital anomalies of the mouth and palate,
  * Those with metabolic (e.g. NEC) and genetic (e.g. osteogenesis imperfecta) diseases,
  * Painful intervention was performed at least 30 minutes before the procedure, Preterm babies will be excluded from the research.

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
OG catheter-related pain | 2 minutes before the OG tube insertion, during the OG tube insertion, 2 minutes after the OG tube insertion
  Neonatal Infant Pain Scale (NIPS): The Newborn Infant Pain Scale (NIPS) was developed by Lawrence et al. in 1993. Turkish validity and reliability were established by Akdovan in 1999. Reliability values were found to be 0.83, 0.83, and 0.86 before, during, and after the procedure, respectively. The newborn infant pain scale is a Likert-type scale consisting of 6 parameters, facial movements (0; relaxed, 1; restless), crying (0; no crying, 1; groaning, 2; loud crying), breathing (0; comfortable, 1; variable-irregular), arm (0: relaxed-free, 1; flexion-extension), leg (0; comfortable-free, 1; flexion-extension) and sleep-wake (0; sleeping-waking peaceful, 1; restless).
OG catheter-related comfort | 2 minutes before the OG tube insertion, during the OG tube insertion, 2 minutes after the OG tube insertion
  The Newborn Comfort Behavior Scale: The newborn comfort behavior scale is a Likert-type scale developed to evaluate the comfort needs, pain, and distress of newborn babies. This scale was developed by Ambuel et al. (1992) to evaluate the comfort, pain, and stress status of newborn babies receiving mechanical ventilator support in the intensive care unit. This scale consists of six parameters: alertness, agitation, respiratory response/crying, body movements, facial tension, and muscle tone. Each item on the scale is scored between 1-5. If the total score obtained as a result of the evaluation is below 13, it is emphasized that the baby is comfortable, if it is 14 and above, the baby's comfort level is low, and additional interventions to increase comfort may be required.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Güven, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No